CLINICAL TRIAL: NCT03549364
Title: A Pilot Study of the Myocardial Effects of an Endurance Race as Evaluated by Computer Tomography
Brief Title: Pilot Study of Myocardial Effects Following an Endurance Race
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, MD PhD professor head of internal medicine, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/429-31
Record Dates: First submitted 2018-05-11; First posted 2018-06-08 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Blood Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endurance race (Experimental): 1. baseline investigations with CT and lab tests
  2. the same CT and lab tests < 24h after an endurance race
  3. CT and lab tests again about 1-2weeks after the race
  Interventions: Behavioral: Endurance Race

INTERVENTIONS:
Behavioral: Endurance Race — 1 CT and lab tests, 2 CT and lab tests within 24h of a race, 3 follow up investigations 1-2 weeks after the race with CT and lab tests

SUMMARY:
Ten healthy subjects perform a baseline computer tomography (CT) of the heart and routine laboratory blood tests for myocardial injury and inflammation.

The same data are collected <24 hours after an endurance race corresponding to a maraton run (i.e. about 40 km of running and/or about 2.5 hours hard training or more). A third collection of lab tests and CT is done a couple of weeks after the race. Magnetic resonance imaging is also performed in parallell to the CT on occasions 2 and 3 in most subjects, serving as a reference for determination of myocardial blood flow.

DETAILED DESCRIPTION:
Ten healthy subjects perform a baseline computer tomography (CT) of the heart and routine laboratory blood tests (troponin T, hs-CRP, CK-mb etc) for myocardial injury and inflammation.

The same data are collected <24 hours after an endurance race corresponding to a maraton run (i.e. about 40 km of running and/or about 2.5 hours hard training or more). A third collection of lab tests and CT is done a couple of weeks after the race. Magnetic resonance imaging (MRI) is also performed in parallell to the CT on occasions 2 and 3 in most subjects, serving as a reference for determination of myocardial blood flow. The CT of the heart includes contrast injection and blood flow will be determined by a recently developed based on very powerful computers using "machine learning".

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects, experienced in long distance running

Exclusion Criteria:

Significant renal, kidney, heart, liver or musculoskeletal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial blood flow by the race? | All investigations are performed < 2 months
  Detection of potential differences in blood flow between occasion 1 and 2 and 3

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No